CLINICAL TRIAL: NCT05827978
Title: A Phase 3, Randomized, Stratified, Observer-Blind, Active-Controlled Study to Evaluate the Immunogenicity, Reactogenicity and Safety of mRNA-1010 Seasonal Influenza Vaccine in Adults 18 Years and Older
Brief Title: Study of mRNA-1010 Seasonal Influenza Vaccine in Adults
Acronym: IGNITE P303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mRNA-1010-P303
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Seasonal Influenza
Keywords: mRNA-1010; Virus Diseases; Flu; Influenza vaccine; Moderna; mRNA vaccine
MeSH Terms: conditions — Virus Diseases; Influenza, Human | interventions — mRNA-1010 influenza vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1010 (Experimental): Participants will receive a single dose of mRNA-1010 by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1010
- Licensed Quadrivalent Inactivated Seasonal Influenza Vaccine (Active Comparator): Participants will receive a single dose of licensed quadrivalent inactivated seasonal influenza vaccine by IM injection on Day 1.
  Interventions: Biological: Licensed Quadrivalent Inactivated Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: mRNA-1010 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1010
Biological: Licensed Quadrivalent Inactivated Seasonal Influenza Vaccine — Sterile suspension for injection
  Other Names: Fluarix Quadrivalent; Fluzone HD
  Arms: Licensed Quadrivalent Inactivated Seasonal Influenza Vaccine

SUMMARY:
This study includes 3 parts: Parts A, B, and C. The purpose of this study is to evaluate the immunogenicity and safety of mRNA-1010 seasonal influenza vaccine in adults.

ELIGIBILITY:
Inclusion Criteria:

* Investigator has assessed that the participant understands and is willing and physically able to comply with protocol mandated follow up, including all procedures.
* For assigned females at birth and of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, and agreement to continue adequate contraception through 90 days following vaccine administration.

Part A:

* At least 18 years of age inclusive, at the time of signing the informed consent form (ICF).

Part B:

* At least 18 and <65 years of age, at the time of signing the ICF.

Part C:

* At least 65 years of age or older, at the time of signing the ICF.

Exclusion Criteria:

* Participant has had close contact with someone with laboratory-confirmed influenza infection or with someone who has been treated with antiviral therapies for influenza (for example, Tamiflu®) within the past 5 days prior to Day 1.
* Participant is acutely ill or febrile (temperature ≥38.0℃elcius [100.4°Fahrenheit]) 72 hours prior to or at the Screening visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day screening window.
* Participant has a history of a diagnosis or condition that, in the judgment of the investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Reported history of congenital or acquired immunodeficiency, immunosuppressive condition or immune-mediated disease, asplenia, or recurrent severe infections.
* Participant has tested positive for influenza by local health authority-approved testing methods within 150 days (for Part A) or 180 days (for Parts B and C) prior to Day 1.
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of mRNA vaccines or any components of the mRNA-1010 or influenza vaccines, including egg protein.
* Participant has received systemic immunosuppressants for >14 days in total within 180 days prior to Day 1 (for corticosteroids, ≥10 mg/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study. Inhaled, nasal and topical steroids are allowed. Intra-articular and epidural steroid injections are not allowed within 28 days before and/or after study intervention dosing.
* Participant has received any vaccine authorized or approved by local health agency ≤28 days prior to study intervention dosing (Day 1) or plans to receive a vaccine authorized or approved by local health agency within 28 days before or after study intervention dosing.
* Participant has received a licensed seasonal influenza vaccine within 5 months (150 days) (for part A) or within 6 months (180 days) (for Parts B and C) prior to Day 1.
* Participant has participated in any investigational seasonal influenza vaccine study within12 months prior to Day 1.
* Participant is not aware whether they have received an influenza vaccine in the most recent influenza season (in the prior 12 months) (for Part A) or since September 2022 (for Parts B and C).
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to Day 1 or plans to donate blood products during the study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8411 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (103):
  - Pinnacle Research Group, Anniston, Alabama
  - North Alabama Research Center LLC, Athens, Alabama
  - Cullman Research Center, Cullman, Alabama
  - Medical Affiliated Research Center Inc, Huntsville, Alabama
  - Desert Clinical Research - CCT, Mesa, Arizona
  - Foothills Research Center - CCT, Phoenix, Arizona
  - Fiel Family & Sports Medicine - PC - CCT, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Velocity Clinical Research, Banning, Banning, California
  - Synexus Clinical Research US, Inc. - Cerritos, Cerritos, California
  - Marvel Clinical Research 002, LLC, Huntington Beach, California
  - Velocity Clinical Research, La Mesa, California
  - Pasadena Clinical Trials, Pasadena, California
  - Artemis Institute For Clinical Research LLC - Riverside - Headlands, Riverside, California
  - Peninsula Research Associates - CRN, Rolling Hills Estates, California
  - Optimal Research, LLC, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - Chase Medical Research LLC - Waterbury, Waterbury, Connecticut
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - NeoClinical Reseaarch, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness Inc, Jupiter, Florida
  - Wr-Msra, Llc., Lake City, Florida
  - Sandhill Research, LLC d/b/a Accel Research Sites Network, Lake Mary, Florida
  - Sandhill Research, LLC d/b/a Accel Research Sites, Lake Mary, Florida
  - University Clinical Research-DeLand, LLC d/b/a Accel Research, Lake Mary, Florida
  - South Florida Research Center, Inc, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Innovation Medical Group, LLC., Palmetto Bay, Florida
  - Suncoast Research Associates, LLC, Pembroke Pines, Florida
  - St. Johns Center for Clinical Research - ERN, Saint Augustine, Florida
  - New Tampa Health, Inc., Tampa, Florida
  - Synexus Clinical Research US, Inc. - The Villages, The Villages, Florida
  - Synexus Clinical Research US, Inc. - Atlanta, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Javara, Inc., Fayetteville, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - CRA, Headlands LLC, Stockbridge, Georgia
  - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials- Ravenswood, Chicago, Illinois
  - DM Clinical Research, River Forest, Illinois
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Velocity Clinical Research, Inc., Overland Park, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Velocity Clinic Research, Inc., Baton Rouge, Louisiana
  - Velocity Clinical Research, Covington, Covington, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Javara Inc., Annapolis, Maryland
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - Oakland Medical Research, Troy, Michigan
  - Clinical Research Institute, Inc - CRN, Minneapolis, Minnesota
  - DelRicht Research, Gulfport, Mississippi
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Methodist Physicians Clinic - CCT Research, Fremont, Nebraska
  - Velocity Clinical Research- Grand Island, Grand Island, Nebraska
  - Velocity Clinical Research (Norfolk - Nebraska) - PPDS, Norfolk, Nebraska
  - Velocity Clinical Research (Omaha - Nebraska) - PPDS, Omaha, Nebraska
  - Velocity Clinical Research, Inc., Omaha, Nebraska
  - Midwest Regional Health Services - LLC - CCT, Omaha, Nebraska
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Velocity Clinical Research (Binghamton - New York) - PPDS, Binghamton, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Velocity Clinical Research, Inc., Vestal, New York
  - Javara Inc., Charlotte, North Carolina
  - Lucas Research Inc., Morehead City, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research, Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research, Inc., Cincinnati, Ohio
  - DelRicht Research, Tulsa, Oklahoma
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - DM Clinical Research - Philadelphia - ERN, Philadelphia, Pennsylvania
  - Velocity Clinical Research - Columbia, Columbia, South Carolina
  - Velocity Clinical Research - Gaffney, Gaffney, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - DelRicht Research, Hendersonville, Tennessee
  - Tekton Research - Austin - PPDS, Austin, Texas
  - Tekton Research, LLC., Beaumont, Texas
  - Javara Inc., Conroe, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - DM Clinical Research, Houston, Texas
  - DM Clinical Research, Humble, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - DM Clinical Research, Sugar Land, Texas
  - Javara Inc., Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - Cope Family Medicine - CCT, Bountiful, Utah
  - J. Lewis Research, Inc., Foothill Family Clinic, Salt Lake City, Utah
  - Olympus Family Medicine - CCT Research, Salt Lake City, Utah
  - South Ogden Family Medicine Ogden Clinic/CCT Research, South Ogden, Utah
  - Clinical Research Partners LLC - Richmond - ERN, Richmond, Virginia

REFERENCES:
- [Result] Soens M, Ananworanich J, Hicks B, Lucas KJ, Cardona J, Sher L, Livermore G, Schaefers K, Henry C, Choi A, Avanesov A, Chen R, Du E, Pucci A, Das R, Miller J, Nachbagauer R. A phase 3 randomized safety and immunogenicity trial of mRNA-1010 seasonal influenza vaccine in adults. Vaccine. 2025 Mar 19;50:126847. doi: 10.1016/j.vaccine.2025.126847. Epub 2025 Feb 7. PMID 39919447
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217501&parentIdentifier=mRNA-1010-P303&attachmentIdentifier=9b318591-af2c-4469-afb9-4a18e6eeb09e&fileName=1010-P303_Temp-0080_Protocol_Template_for_Registrations_19Jan23.docx&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Fluarix Quadrivalent Influenza Vaccine (QIV): Participants received a single dose of Fluarix QIV by intramuscular (IM) injection on Day 1.
- Part A: mRNA-1010; Part B: mRNA-1010; Part C: mRNA-1010: Participants received a single dose of mRNA-1010 by IM injection on Day 1.
- Part B: Fluarix QIV: Participants received a single dose of Fluarix QIV by IM injection on Day 1.
- Part C: Fluzone High Dose (HD) QIV: Participants received a single dose of Fluzone HD QIV by IM injection on Day 1.
Period: Overall Study
Arm/Group | Part A: Fluarix Quadrivalent Influenza Vaccine (QIV) | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone High Dose (HD) QIV | Part C: mRNA-1010
Started | 1189 | 1225 | 1494 | 1500 | 1496 | 1507
Safety Set (All randomized participants who received any study intervention. Participants were included in the group corresponding to the study intervention that they actually received.) | 1180 | 1220 | 1488 | 1492 | 1490 | 1502
Completed | 1106 | 1113 | 1425 | 1434 | 1456 | 1484
Not Completed | 83 | 112 | 69 | 66 | 40 | 23
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 1 | 5 | 2 | 3 | 1 | 3
Not completed — Lost to Follow-up | 57 | 88 | 54 | 47 | 25 | 10
Not completed — Noncompliance with Study Procedures | 0 | 1 | 1 | 1 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 1 | 2 | 1 | 1
Not completed — Protocol Violation | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 16 | 10 | 12 | 10 | 9
Not completed — Other Than Specified | 0 | 0 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomization set included all participants who were randomly assigned to the study intervention, regardless of the participants' study intervention status in the study. Participants were analyzed according to the group to which they were randomized.
Groups:
- Part A: Fluarix QIV; Part B: Fluarix QIV: Participants received a single dose of Fluarix QIV by IM injection on Day 1.
- Part C: Fluzone HD QIV: Participants received a single dose of Fluzone HD QIV by IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010 | Total
Number analyzed (Participants) | 1189 | 1225 | 1494 | 1500 | 1496 | 1507 | 8411
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 919 | 951 | 1494 | 1500 | 1 | 0 | 4865
  >=65 years | 270 | 274 | 0 | 0 | 1495 | 1507 | 3546
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 627 | 663 | 906 | 882 | 855 | 883 | 4816
  Male | 562 | 562 | 588 | 618 | 641 | 624 | 3595
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 226 | 262 | 392 | 406 | 456 | 451 | 2193
  Not Hispanic or Latino | 948 | 941 | 1083 | 1076 | 1025 | 1041 | 6114
  Unknown or Not Reported | 15 | 22 | 19 | 18 | 15 | 15 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 856 | 922 | 970 | 1020 | 1224 | 1257 | 6249
  Race: Black or African American | 274 | 250 | 446 | 420 | 237 | 227 | 1854
  Race: Asian | 34 | 27 | 28 | 24 | 10 | 10 | 133
  Race: American Indian or Alaska Native | 5 | 7 | 12 | 12 | 9 | 4 | 49
  Race: Native Hawaiian or Other Pacific Islander | 1 | 3 | 4 | 4 | 0 | 2 | 14
  Race: Multiple | 11 | 11 | 18 | 6 | 6 | 2 | 54
  Race: Other | 3 | 3 | 7 | 11 | 4 | 1 | 29
  Race: Not Reported | 3 | 0 | 6 | 2 | 2 | 3 | 16
  Race: Unknown | 2 | 2 | 3 | 1 | 4 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibody Levels as Measured by Hemagglutination Inhibition (HAI)
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria and Yamagata strains. Antibody values reported as below lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Values greater than the upper limit of quantification (ULOQ) were converted to the ULOQ.
Time Frame: Day 29
Population: The Per-Protocol Immunogenicity Set (PPIS) included all randomized participants who received the planned dose of study intervention, complied with the immunogenicity testing schedule for Baseline and Day 29, and had no significant protocol deviations that impacted key or critical data. Participants were analyzed according to the group to which they were randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1135 | 1185 | 1426 | 1441 | 1409 | 1425
titer
  Influenza A H1N1 Antibody | 147.49 [138.07 to 157.55] | 220.17 [207.30 to 233.84] | 137.90 [129.89 to 146.40] | 208.10 [196.43 to 220.47] | 130.09 [122.86 to 137.74] | 174.81 [165.15 to 185.04]
  Influenza A H3N2 Antibody | 107.21 [101.11 to 113.68] | 152.56 [144.13 to 161.48] | 97.18 [91.74 to 102.95] | 157.88 [148.45 to 167.91] | 116.24 [109.47 to 123.44] | 141.62 [133.29 to 150.46]
  Influenza B/Victoria Antibody | 155.94 [147.78 to 164.55] | 198.55 [188.44 to 209.22] | 150.90 [144.37 to 157.73] | 196.71 [187.68 to 206.17] | 195.97 [187.44 to 204.89] | 248.03 [237.34 to 259.21]
  Influenza B/Yamagata Antibody | 146.63 [138.91 to 154.78] | 182.94 [173.61 to 192.76] | 113.76 [109.21 to 118.51] | 158.58 [151.55 to 165.93] | 91.94 [88.33 to 95.71] | 104.82 [100.70 to 109.11]

2. Primary Outcome: Percentage of Participants Reaching Seroconversion, as Measured by HAI
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria and Yamagata strains. Seroconversion rate was defined as the percentage of participants with either a Baseline HAI titer <1:10 and a postbaseline titer ≥1:40 or a Baseline HAI titer ≥1:10 and a minimum 4-fold rise in postbaseline HAI antibody titer. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were converted to the ULOQ.
Time Frame: Day 29
Population: The PPIS included all randomized participants who received the planned dose of study intervention, complied with the immunogenicity testing schedule for Baseline and Day 29, and had no significant protocol deviations that impacted key or critical data. Participants were analyzed according to the group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1135 | 1185 | 1426 | 1441 | 1409 | 1425
percentage of participants
  Influenza A H1N1 Antibody | 34.9 [32.12 to 37.74] | 50.2 [47.32 to 53.10] | 45.0 [42.42 to 47.65] | 64.4 [61.87 to 66.88] | 36.3 [33.75 to 38.84] | 49.7 [47.06 to 52.31]
  Influenza A H3N2 Antibody | 32.2 [29.45 to 34.96] | 51.1 [48.17 to 53.94] | 44.0 [41.37 to 46.59] | 66.4 [63.91 to 68.85] | 47.8 [45.20 to 50.48] | 56.4 [53.80 to 59.02]
  Influenza B/Victoria Antibody | 17.0 [14.86 to 19.32] | 26.6 [24.09 to 29.20] | 18.4 [16.39 to 20.48] | 33.0 [30.54 to 35.46] | 20.2 [18.09 to 22.35] | 29.8 [27.46 to 32.27]
  Influenza B/Yamagata Antibody | 24.7 [22.19 to 27.29] | 33.2 [30.57 to 36.01] | 23.4 [21.25 to 25.71] | 35.6 [33.12 to 38.13] | 20.2 [18.09 to 22.35] | 26.0 [23.77 to 28.40]

3. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs, representative of vaccine reactogenicity, were collected in an electronic diary (eDiary). Local ARs: injection site pain, erythema (redness), swelling/induration (hardness); and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Per prespecified analysis, only solicited ARs that were assessed and confirmed by the Investigator as both serious and related to IP were recorded as an adverse event. These adverse events were recorded as a serious AE (SAE) and are included in the summary of SAEs in the "Reported Adverse Events" section.
Time Frame: Up to 7 days after study injection
Population: Solicited Safety Set included all randomized participants who received any study intervention and contributed any solicited AR data. Participants were included in the group corresponding to the study intervention that they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1180 | 1220 | 1488 | 1492 | 1490 | 1502
Participants | 682 | 1060 | 796 | 1158 | 734 | 1131

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Unsolicited AEs included any AE not collected as a solicited AR, and also included solicited ARs assessed and confirmed as both serious and related by the Investigator. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Up to 28 days after study injection
Population: Safety Set included all randomized participants who received any study intervention. Participants were included in the group corresponding to the study intervention that they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1180 | 1220 | 1488 | 1492 | 1490 | 1502
Participants | 134 | 145 | 134 | 147 | 137 | 155

5. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs), SAEs, and AEs Leading to Discontinuation
Description: An MAAE was an AE that led to an unscheduled visit to a healthcare practitioner. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required. An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability, was a congenital anomaly/birth defect, or was an important medical event. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 181
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1180 | 1220 | 1488 | 1492 | 1490 | 1502
Participants
  MAAEs | 195 | 226 | 223 | 217 | 248 | 257
  AESIs | 2 | 1 | 0 | 1 | 1 | 2
  SAEs | 21 | 27 | 22 | 25 | 38 | 41
  AEs Leading to Discontinuation | 1 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Percentage of Participants With HAI Titer ≥1:40
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria and Yamagata strains.
Time Frame: Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1135 | 1185 | 1426 | 1441 | 1409 | 1425
percentage of participants
  Influenza A H1N1 Antibody | 93.7 [92.17 to 95.08] | 96.7 [95.53 to 97.65] | 92.0 [90.47 to 93.36] | 96.4 [95.29 to 97.29] | 92.3 [90.82 to 93.67] | 96.5 [95.40 to 97.38]
  Influenza A H3N2 Antibody | 92.0 [90.25 to 93.50] | 97.0 [95.92 to 97.93] | 86.4 [84.51 to 88.13] | 92.6 [91.17 to 93.94] | 88.9 [87.10 to 90.45] | 92.8 [91.38 to 94.13]
  Influenza B/Victoria Antibody | 99.3 [98.62 to 99.70] | 99.7 [99.14 to 99.91] | 99.4 [98.90 to 99.76] | 99.4 [98.82 to 99.71] | 99.5 [98.98 to 99.80] | 100 [99.74 to 100.00]
  Influenza B/Yamagata Antibody | 97.5 [96.45 to 98.35] | 98.5 [97.61 to 99.10] | 97.4 [96.44 to 98.17] | 97.8 [96.88 to 98.48] | 93.7 [92.28 to 94.90] | 96.1 [95.01 to 97.08]

7. Secondary Outcome: Geometric Mean Fold-Rise (GMFR) of Postinjection Anti-HA Antibodies for Influenza, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria and Yamagata strains. The GMFR measured the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% confidence interval (CI) for GMFR was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Baseline (Day 1) to Day 29
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1135 | 1185 | 1426 | 1441 | 1409 | 1425
ratio
  Influenza A H1N1 Antibody | 2.78 [2.59 to 2.99] | 4.03 [3.80 to 4.27] | 3.29 [3.10 to 3.49] | 4.99 [4.73 to 5.26] | 2.60 [2.47 to 2.74] | 3.49 [3.32 to 3.67]
  Influenza A H3N2 Antibody | 2.60 [2.46 to 2.76] | 3.68 [3.49 to 3.87] | 3.16 [2.99 to 3.35] | 5.33 [5.04 to 5.64] | 3.40 [3.22 to 3.60] | 4.12 [3.90 to 4.36]
  Influenza B/Victoria Antibody | 1.75 [1.67 to 1.84] | 2.22 [2.12 to 2.32] | 1.85 [1.78 to 1.93] | 2.47 [2.37 to 2.57] | 1.89 [1.82 to 1.97] | 2.35 [2.26 to 2.45]
  Influenza B/Yamagata Antibody | 2.10 [1.99 to 2.22] | 2.63 [2.52 to 2.76] | 2.01 [1.93 to 2.10] | 2.79 [2.67 to 2.91] | 1.92 [1.85 to 2.00] | 2.20 [2.13 to 2.28]

8. Other Pre Specified Outcome: Number of Deaths Related to Study Drug
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, whether or not it was considered related to study drug. The investigator assessed causality (that is, whether there is a reasonable possibility that the study drug caused the death). The relationship was characterized using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable AND/OR the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable. The death was more likely explained by the study drug than by another cause.
Time Frame: Day 1 through Day 181
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
Number analyzed (Participants) | 1189 | 1225 | 1494 | 1500 | 1496 | 1507
Participants
  Number of deaths | 1 | 5 | 2 | 3 | 1 | 3
  Number of deaths assessed by Sponsor as related to study drug | 0 | 0 | 0 | 0 | 0 | 0
  Number of deaths assessed by Investigator as related to study drug | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were collected from Day 1 through Day 181. Other (not including serious) unsolicited adverse events were collected up to 28 days after study injection (that is, Day 1 up to Day 29)
Description: The all-cause mortality was based on the randomization set. The serious and other (not including serious) adverse events were based on the safety set which consisted of all randomized participants who received any study intervention. Participants were included in the group corresponding to the study intervention that they actually received.
Arm/Group | Part A: Fluarix QIV | Part A: mRNA-1010 | Part B: Fluarix QIV | Part B: mRNA-1010 | Part C: Fluzone HD QIV | Part C: mRNA-1010
All-Cause Mortality (participants affected / at risk) | 1/1189 | 5/1225 | 2/1494 | 3/1500 | 1/1496 | 3/1507
Serious Adverse Events (participants affected / at risk) | 21/1180 | 27/1220 | 22/1488 | 25/1492 | 38/1490 | 41/1502
Other Adverse Events (participants affected / at risk) | 0/1180 | 0/1220 | 0/1488 | 0/1492 | 0/1490 | 0/1502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Fluarix QIV (N=1180) | Part A: mRNA-1010 (N=1220) | Part B: Fluarix QIV (N=1488) | Part B: mRNA-1010 (N=1492) | Part C: Fluzone HD QIV (N=1490) | Part C: mRNA-1010 (N=1502)
Abortion infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral cavernous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT05827978/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT05827978/SAP_001.pdf